CLINICAL TRIAL: NCT00620932
Title: Feasibility of Endurance Exercise Training on Cardiovascular Risk Factors Following Radical Prostatectomy Among Men With Localized Prostate Cancer; A Community-Based Intervention
Brief Title: Exercise Training Among Men With Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00002501
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Prostatectomy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): These patients will continue with whatever routine exercise they already engage in.
- Exercise Arm (Experimental): These patients will participate in a controlled, supervised exercise program.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Patients will be randomly assigned to groups and will either be given an exercise program individually tailored to them for them to participate in for 6 months or else be wait-listed for 6 months and remain on whatever exercise regimen they were already on.
  Arms: Exercise Arm

SUMMARY:
The primary objective is to determine the feasibility and acceptability of a home-based endurance exercise program among men diagnosed with clinically localized prostate cancer.

DETAILED DESCRIPTION:
Approximately 40 people will take part in this study and all of these people will take part at Duke University Medical Center.

Participation in this study involves the following.

* We will ask you to perform a cardiopulmonary exercise test (walking stress test) to determine if you have any undiagnosed cardiovascular health problems that may limit your ability to participate in an exercise training program. This test will take place at the Duke Center for Living on Duke University Campus.
* Complete a body composition assessment. This test is designed to determine your body fat and lean body tissue (muscle mass) percentage and will consist of you sitting quietly in a chamber with appropriate medical supervision. This test also will take place at the Duke Center for Living on Duke University Campus.
* Complete two questionnaires one at the beginning and one at the end that asks about how you are feeling and about your physical activity levels. The questionnaire takes about 20-30 minutes.
* Provide two blood samples one at the beginning and one at the end to measure levels of cardiovascular disease risk factors (cholesterol levels, c-reactive protein and insulin levels) in your blood that may be influenced by exercise. Blood collection will be drawn by medical staff at Duke University. The amount of blood drawn is approximately 2 teaspoons (10ml).
* We will also collect information on how much treatment you receive as well as how many and what type of side-effects you have from your medical treatment. This information will be obtained from your medical chart following the completion of your treatment.

Following the successful completion of all initial tests and procedures (as described above), you will be randomly assigned (like flipping a coin) to one of the following two groups:

1. Exercise Training Group: You will be given a customized training program aimed at increasing cardiorespiratory fitness. You will be asked to exercise 3 to 5 times per week. All sessions will include a 5 minute warm-up and 5 minute cool-down at the beginning and end of each session totaling 30-45 minutes per session. You will also receive a heart rate monitor to record each exercise session to monitor adherence and compliance. You will receive telephone calls every two weeks to provide encouragement, outline goals, and provide feedback on study progress.

   OR
2. Wait-List Control Group: You will be asked to maintain your usual exercise levels during the 6 month study period. You will receive telephone calls to report your levels of exercise during the study. After study completion you will receive a heart rate monitor and an individualized exercise prescription based on your cardiorespiratory fitness test at the end of the study period (6 months).

ELIGIBILITY:
Inclusion Criteria:

1. Legal age (>18 years old)
2. An interval of at least 6 weeks between prior radical prostatectomy and study enrollment
3. Karnofsky performance status of at least 70% at study entry
4. Estimated life expectancy of ≥6 months
5. Ability to read and understand English
6. Attending urologist approval
7. Signed informed consent
8. Willingness to be randomized; and
9. No contraindications to exercise as recommended by the American Thoracic Society

Exclusion Criteria:

1. Acute myocardial infarction (6 weeks)
2. Unstable angina
3. Uncontrolled arrhythmias causing symptoms or hemodynamic compromise
4. Syncope
5. Acute endocarditis
6. Acute myocarditis or pericarditis
7. Uncontrolled heart failure
8. Acute pulmonary embolus or pulmonary infarction
9. Thrombosis of lower extremities
10. Suspected dissecting aneurysm
11. Uncontrolled asthma
12. Pulmonary edema
13. Room air desaturation at rest ≤85%
14. Respiratory failure
15. Acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise; and
16. Mental impairment leading to inability to cooperate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness will be determined using a incremental treadmill test with 12-lead ECG monitoring. | 6 months

SECONDARY OUTCOMES:
Fasting lipids will be assessed. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jones, PHd, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Jones LW, Hornsby WE, Freedland SJ, Lane A, West MJ, Moul JW, Ferrandino MN, Allen JD, Kenjale AA, Thomas SM, Herndon JE 2nd, Koontz BF, Chan JM, Khouri MG, Douglas PS, Eves ND. Effects of nonlinear aerobic training on erectile dysfunction and cardiovascular function following radical prostatectomy for clinically localized prostate cancer. Eur Urol. 2014 May;65(5):852-5. doi: 10.1016/j.eururo.2013.11.009. Epub 2013 Nov 22. PMID 24315706
- See also: Preston Robert Tisch Brain Tumor Center at Duke — http://www.cancer.duke.edu/btc/